CLINICAL TRIAL: NCT03567590
Title: A Prospective, Multicentre, Randomized, Controlled, Blinded-endpoint Study to Evaluate the Efficacy and Safety of Sphenopalatine Ganglion Pulsed Radiofrequency Treatment for Cluster Headache
Brief Title: The Efficacy and Safety of Sphenopalatine Ganglion Pulsed Radiofrequency Treatment for Cluster Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Sanbo Brain Hospital (Other); Jilin Province People's Hospital (Unknown)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY 2018-027-02
Record Dates: First submitted 2018-05-22; First posted 2018-06-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Cluster Headache
Keywords: Cluster Headache, pulsed radiofrequency
MeSH Terms: conditions — Cluster Headache | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulsed Radiofrequency Group (Experimental): This group will undergo pulsed radiofrequency treatment.
  Interventions: Procedure: Pulsed Radiofrequency treatment
- Nerve Block Group (Active Comparator): This group will undergo nerve block treatment.
  Interventions: Procedure: Nerve Block treatment

INTERVENTIONS:
Procedure: Pulsed Radiofrequency treatment — The pulse treatment generator (PMF-21-100-5, Baylis Medical Inc., Montreal, Canada) with a length of 10 cm, 21-gauge, and an active tip length of 5 mm is inserted vertically into the puncture point. The pulse treatment generator is set to the pulsed radiofrequency automatic mode, with a temperature of 42 °C, pulse frequency of 2 Hz, pulse width of 20 ms, and treatment duration of 360s.
  Arms: Pulsed Radiofrequency Group
Procedure: Nerve Block treatment — A mixture of 40 mg Triamcinolone + 2 ml of 1% Bupivacaine + 2 ml of 2% mepivacaine + 1:100000 epinephrine is injected for nerve block treatment using a puncture needle.
  Arms: Nerve Block Group

SUMMARY:
The investigators aim to investigate the effectiveness and safety of sphenopalatine ganglion pulsed radiofrequency on cluster headache.

DETAILED DESCRIPTION:
The investigators aim to investigate whether the sphenopalatine ganglion pulsed radiofrequency treatment is better than traditional sphenopalatine ganglion nerve block technology and provides medical evidence for the clinical application and promotion of sphenopalatine ganglion pulsed radiofrequency treatment to provide a minimally invasive, safe, and effective treatment for patients with cluster headache who do not respond to drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cluster headache is confirmed according to the diagnostic criteria of the 2018 International Classification of Headache Disorders 3rd edition (ICHD-3);
* patient's age is between 18 and 60 years;
* patients seek treatment in the pain clinics of hospitals participating in the study within 5 days of the onset of the cluster period; pain conditions of patients remain the same after conservative treatment of conventional oral medication, or the reduction rates are less than 50% in pain degree during headache attacks, headache attack frequency, duration of each headache attack, and auxiliary analgesic drug dosage; and
* patients signed the informed consent.

Exclusion Criteria:

* abnormalities in blood measurements, liver and kidney function, blood glucose, coagulation, electrocardiogram, and chest radiograph;
* infection at the puncture site;
* previous mental illness;
* previous history of narcotic drug abuse;
* history of anticoagulant and antiplatelet aggregation drugs;
* implantable pulse generator;
* previous history of invasive treatments such as sphenopalatine ganglion radiofrequency thermocoagulation and chemical destruction;
* pregnant or breastfeeding patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Duration of the cluster period | Within 1 year (the cluster period is not over 3 months generally)
  The duration of the cluster period is defined as the total duration of the headache, including the pain attack time before and after treatment.

SECONDARY OUTCOMES:
The degree of pain during headache attacks after treatment | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 1 year after surgery
  Evaluated by numeric rating scale (NRS, 0 points for no pain and 10 points for the most severe pain)
Headache attack frequency | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 1 year after surgery
  The number of attacks per day
Duration of each headache attack | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 1 year after surgery
  Duration of each headache attack after treatment
Dose of auxiliary analgesic drugs | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 1 year after surgery
  Dose of auxiliary analgesic drugs per day
Duration of remission period | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 1 year after surgery
  From the end of this cluster period to the beginning of the next cluster period
Patient satisfaction | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 1 year after surgery
  Patient satisfactory scale (PSS) evaluation (0 for unsatisfactory, and 10 for very satisfied).
Effective rate | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, and 1 year after surgery
  The effectiveness rate is calculated as follows: effectiveness rate = the number of effective patients / total number of patients in this group × 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (3):
- China (3):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing Sanbo Brain Hospital, Beijing, Beijing Municipality
  - Jilin Province People's Hospital, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weaver-Agostoni J. Cluster headache. Am Fam Physician. 2013 Jul 15;88(2):122-8. PMID 23939643
- [Background] Penarrocha-Diago M, Boronat A, Penarrocha-Oltra D, Ata-Ali J, Bagan JV, Penarrocha-Diago M. Clinical course of patients with episodic cluster headache treated with corticosteroids inproximity to the sphenopalatine ganglion: a preliminary study of 23 patients. Med Oral Patol Oral Cir Bucal. 2012 May 1;17(3):e477-82. doi: 10.4317/medoral.17578. PMID 22143727
- [Background] Lepper A, Frese A, Summ O, Nofer JR, Evers S. Hypothalamic dopaminergic stimulation in cluster headache. Cephalalgia. 2013 Oct;33(14):1155-9. doi: 10.1177/0333102413487445. Epub 2013 Apr 29. PMID 23630400
- [Background] Loomba V, Upadhyay A, Kaveeshvar H. Radiofrequency Ablation of the Sphenopalatine Ganglion Using Cone Beam Computed Tomography for Intractable Cluster Headache. Pain Physician. 2016 Sep-Oct;19(7):E1093-6. PMID 27676681
- [Background] Kohlmeier C, Behrens P, Boger A, Ramachandran B, Caparso A, Schulze D, Stude P, Heiland M, Assaf AT. Improved surgical procedure using intraoperative navigation for the implantation of the SPG microstimulator in patients with chronic cluster headache. Int J Comput Assist Radiol Surg. 2017 Dec;12(12):2119-2128. doi: 10.1007/s11548-016-1512-2. Epub 2017 Jan 12. PMID 28083804
- [Background] Barloese MC, Jurgens TP, May A, Lainez JM, Schoenen J, Gaul C, Goodman AM, Caparso A, Jensen RH. Cluster headache attack remission with sphenopalatine ganglion stimulation: experiences in chronic cluster headache patients through 24 months. J Headache Pain. 2016 Dec;17(1):67. doi: 10.1186/s10194-016-0658-1. Epub 2016 Jul 26. PMID 27461394
- [Derived] Li J, Ren H, Wang B, Wu D, Luo F. Multicentre, prospective, randomised, controlled, blinded-endpoint study to evaluate the efficacy and safety of pterygopalatine ganglion pulsed radiofrequency treatment for cluster headache: study protocol. BMJ Open. 2019 Mar 23;9(3):e026608. doi: 10.1136/bmjopen-2018-026608. PMID 30904875